CLINICAL TRIAL: NCT03765827
Title: Effect of the Application of Vitamin E Ointment, Over Staple Lines and Anastomosis in Roux-en-Y Gastric Bypass, on Postoperative Pain
Brief Title: Vitamin E on Staple Line and Anastomoses of Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC 18-11
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the epidemiology nurse will not know the treatgment assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin E acetate (Experimental): Vitamin E acetate ointment will be applied over the staple lines and anastomoses in Roux-en-Y gastric bypass
  Interventions: Drug: Vitamine E Acetate
- Control group (Sham Comparator): No ointment will be applied
  Interventions: Drug: No application of vitamin E acetate

INTERVENTIONS:
Drug: Vitamine E Acetate — Vitamin E acetate ointment will be applied over the staple lines and anastomoses in Roux-en-Y gastric bypass
  Other Names: Vitamin E acetate ointment
  Arms: Vitamin E acetate
Drug: No application of vitamin E acetate — Vitamin E acetate ointment will not be applied in this group
  Other Names: No application of vitamin E acetate oinment
  Arms: Control group

SUMMARY:
Patients will be randomized into 2 groups:

* Vit E group: Vitamin E ointment will be applied over staple lines and anastomoses
* Control group: Vitamin E will not be applied

Postoperative pain will be assessed 24 hours after surgery.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* Vit E group: Vitamin E acetate ointment will be applied over staple lines and anastomoses in Roux-en-Y gastric bypass.
* Control group: Vitamin E will not be applied

Postoperative pain will be assessed 24 hours after surgery, by means of visuala analogic scale (ranging from 0 to 100mm).

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 Kg/m2 or >35 Kg/m2 associated to obesity-related comorbidities
* Patients undergoing Roux-en-Y gastric bypass as bariatric procedure
* Patients accepting to participate in the study and signing and Informed Consent form

Exclusion Criteria:

* Patients undergoing other bariatric techniques
* Patients undergoing Roux-en-Y gastric bypass as revisional procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Postoperative pain will be assessed by means of a Visual Analogic Scale, ranging from 0 (absence of pain) to100mm (unbearable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia, MD, PhD, Study Director — Hospital Rey Juan Carlos
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Garcia A, Ferrigni C, Duran M. Application of Vitamin E Acetate on Staple Lines and Anastomoses of Roux-en-Y Gastric Bypass: Impact on Postoperative Pain and Acute Phase Reactants. Obes Surg. 2020 Aug;30(8):2988-2993. doi: 10.1007/s11695-020-04635-9. PMID 32342266